CLINICAL TRIAL: NCT02739490
Title: Effect of the Pelvic Loin Musculature Training on the Dynamic Hip Stabilization: Random Clinical Trial
Brief Title: Effect of the Pelvic Loin Musculature Training on the Dynamic Hip Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Centro-Oeste (Other)
Responsible Party: Principal Investigator, Camila Lazarin Gallina, principal investigator, Universidade Estadual do Centro-Oeste
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CG 001
Record Dates: First submitted 2016-03-11; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Exercise Addiction
Keywords: physiotherapeutic techniques; pelvis; Muscle strength

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group control (No Intervention): It does not perform any kind of guided exercise.
- Core Training Group (Experimental): The training was distributed in four positions defined ventral plank, side plank left, right side board and bridge semiflexion knees, respectively. With time isometric contraction of 30 seconds repeated four times with rest 30 seconds between repetitions. During 10 sessions distributed twice weekly.
  Interventions: Procedure: Core Training Group

INTERVENTIONS:
Procedure: Core Training Group — Performs oriented exercise segmental stabilization lumbar-pelvic.
  Arms: Core Training Group

SUMMARY:
Introduction: The stability of the pelvis is of great importance in body balance as a whole, can be improved by training the pelvic muscles fillet (MLP), which is characterized by low intensity isometric synchronous and the deep muscles of the trunk. This study aims to determine the effect of a stability program target, with the training of the MLP region on pelvic stability.

DETAILED DESCRIPTION:
This study aims to determine the effect of a stability program target, with the training of the MLP region on pelvic stability. Materials and Methods: We recruited 20 volunteers of both sexes were randomly divided into control group (CG) and training group (TG). The evaluations were performed before and after training the MLP. The training was held four isometrics series with a time of 30 seconds with 30 seconds rest in between reps during 10 sessions distributed twice weekly.

ELIGIBILITY:
Inclusion Criteria:

* considered individuals of both sexes, aged 18 and 35
* absence of low back pain
* lack of musculoskeletal dysfunction in the lower limbs
* have never participated in any stabilization training program of the MLP region
* agree to the Terms Informed consent form (ICF) and the sign voluntarily.

Exclusion Criteria:

* the study of abandonment by a participant
* the disagreement with the terms of IC and its not signing
* the volunteer does not understand the implementation of dynamic hip stabilization test
* present cramps or pain during the test and / or training
* historical column in injury, knee and / or ankle.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Values of pelvic tilts , left and right expressed in degrees ( ° ) , the control group (CG ) and training group (TG ) . | 5 weeks
Values of unilateral pelvic tilts between the control group (CG) and training group (TG ) after training. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Camila Gallina, Principal Investigator — Universidade Estadual do Centro-Oeste

IPD SHARING:
Plan to Share IPD: Undecided